CLINICAL TRIAL: NCT06484504
Title: Effect of Kombucha Consumption on the Microbiome in Healthy Subjects
Acronym: KOMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: GT's Living Foods (Unknown)
Responsible Party: Principal Investigator, Jack Gilbert, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 210823
Record Dates: First submitted 2024-06-07; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Health Behavior
Keywords: Microbiome; Inflammation; Biochemical indicators
MeSH Terms: conditions — Health Behavior; Inflammation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention to be administered
- Kombucha group (Experimental): Two servings of a 16 oz commercial kombucha beverage daily for four weeks
  Interventions: Dietary Supplement: Kombucha beverage

INTERVENTIONS:
Dietary Supplement: Kombucha beverage — After 4-weeks of consuming a beige diet (i.e. low-fiber, low polyphenol diet), 20 subjects (kombucha group) will consume one bottle (two servings) of kombucha daily for 4 weeks and 10 subjects (control group) will not change their dietary habits
  Arms: Kombucha group

SUMMARY:
This proposed pilot study will assess the ability of consumption of two servings of kombucha daily to decrease inflammation, alter the gut microbiome composition, and improve intestinal wellbeing in a free-living population. The primary objective is to determine changes in the fecal microbiome composition. Secondary outcomes will be bacterial metabolites (fecal indole propionic acid, calprotectin), serum interleukin (IL) 6, interleukin (IL) 10, C-reactive protein (CRP), C-peptide, insulin, fasting glucose, Homeostatic Model Assessment for Insulin Resistance (HOMA), 14-day continuous glucose monitor, digestive health, dietary information, general Health & Wellness at 4 and 8 weeks.

DETAILED DESCRIPTION:
An altered intestinal gut microbiota, i.e. dysbiosis, has been associated with the development of intestinal disease including inflammatory bowel disease and metabolic diseases such as obesity, type 2 diabetes mellitus (T2DM), and cardiovascular disease. Fermented foods such as Kefir, Kombucha, Miso, and Kimchi contain potentially probiotic microorganisms. The characteristic microbiome in kombucha includes several genera of acetic acid bacteria, yeasts and lactic acid bacteria. Interactions between bacteria and yeast species can lead to the generation of a wide range of metabolites with interesting bioactivities such as organic acids, sugars, phenolic compounds. Kombucha produced from green and black tea contain many phenolic compounds, which contribute to its antioxidant and anti-inflammatory activity and effect on the intestinal microbiota. However, there is a lack of intervention trials investigating the health benefits of fermented foods. Therefore, the investigators propose a human intervention study to assess if daily consumption of two servings of kombucha will alter the intestinal microbiota, decrease inflammation, and improve digestive health in a two-phase design in a free-living population.

This will be a randomized, controlled, two arm intervention study. The study will be conducted in 30 healthy, free-living subjects (21-55 years). After 4-weeks of consuming a beige diet (i.e. low-fiber, low polyphenol diet), 20 subjects will consume one bottle (two servings) of kombucha daily for 4 weeks and 10 subjects will not change their dietary habits. At baseline (week 0), week 4 and 8, blood will be collected. On the day prior to the study visits at week 4 and 8, participants will collect a stool and bring it to the lab. On the day of study visit week 0, 4, and 8, body weight and composition will be determined, and questionnaires and 3-day food record will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Typically consume low fiber/polyphenol diet (beige diet)
* BMI within 25-29.9 kg/m2

Exclusion Criteria:

* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement, which interfere with the absorption of polyphenols
* History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination
* Is unable or unwilling to comply with the study protocol
* Using prebiotics, probiotics, yogurt, and/or any fiber supplements regularly
* Taking antibiotics or laxatives within the past 3 months
* Allergy or sensitivity to kombucha
* In the opinion of the study investigator, any subject who demonstrate a risk of non-compliance with study procedure, or one who cannot read, understand, or complete study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Change in microbiome species richness and abundance of participants at time point 2 (week 8) from baseline (week 0) | Three time points which are baseline(week 0), time point 1(week 4) and time point 2 (week 8)
  Shotgun metagenomic sequencing will be employed on fecal samples collected at three time points in the study period to capture the microbiome profile

SECONDARY OUTCOMES:
Change in fasting blood glucose levels at time point 2 from baseline (week 0) | Baseline (week 0) and time point 2 (week 8)
  fasting glucose (mg/dL) will be measured from blood samples during the study
Change in fasting blood insulin levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0) and time point 2 (week 8)
  Fasting insulin (μU/mL) will be measured from blood samples during the study
Change in fasting blood triglycerides levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0) and time point 2 (week 8)
  Fasting triglycerides (mg/dL) will be measured from blood samples during the study
Change in fasting blood cholesterol levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0) and time point 2 (week 8)
  Total cholesterol, High density lipoprotein (HDL) cholesterol and low density lipoprotein (LDL) cholesterol (mg/dL) will be measured from blood samples during the study
Change in fasting blood glycated hemoglobin (HbA1C) at time point 2 (week 8) from baseline (week 0) | Baseline (week 0) and time point 2 (week 8)
  Glycated hemoglobin (hbA1c) (%) will be measured from blood samples during the study
Change in serum interleukin (IL)10 levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0), time point 1 (week 4) and time point 2 (week 8)
  Measurement of serum interleukin (IL) 10 levels (pg/mL) by flow cytometry
Change in serum interleukin (IL) 6 levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0), time point 1 (week 4) and time point 2 (week 8)
  Measurement of serum interleukin (IL) 6 levels (pg/mL) by flow cytometry
Change in serum C-reactive protein (CRP) levels at time point 2 (week 8) from baseline (week 0) | Baseline (week 0), time point 1 (week 4) and time point 2 (week 8)
  Measurement of serum C-reactive protein (CRP) levels by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Gilbert, Ph.D., Principal Investigator — UC San Diego
Locations (1):
- UC San Diego ACTRI, La Jolla, California, United States